CLINICAL TRIAL: NCT00369070
Title: A Phase 2, Multicenter, Open Label, Randomized Trial of AMG 706 or Bevacizumab in Combination With Paclitaxel and Carboplatin for Advanced Non-squamous Non-small Cell Lung Cancer
Brief Title: A Phase 2 Trial of AMG 706 or Bevacizumab in Combination With Chemo for Advanced NSCLC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20060136
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Last update posted 2018-01-04 (Actual); Status verified 2018-01

CONDITIONS: Advanced Non-squamous NSCLC
Keywords: AMG 706; Bevacizumab; Paclitaxel and Carboplatin; Randomized; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; motesanib diphosphate; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental): AMG 706 125 mg once daily (QD) and paclitaxel and carboplatin chemotherapy regimen (paclitaxel 200 mg/m2 and carboplatin at AUC of 6 mg/mL x min) on day 1 of each 3 week cycle for a maximum of 6 cycles.
  Interventions: Drug: AMG 706; Drug: Paclitaxel; Drug: Carboplatin
- B (Experimental): AMG 706 75 mg twice daily every 12 ± approximately 1 hour for 5 days followed by a 2 day treatment free period every 7 days and paclitaxel and carboplatin chemotherapy regimen (paclitaxel 200 mg/m2 and carboplatin at AUC of 6 mg/mL x min) on day 1 of each 3 week cycle for a maximum of 6 cycles.
  Interventions: Drug: AMG 706; Drug: Paclitaxel; Drug: Carboplatin
- C (Active Comparator): Bevacizumab 15 mg/kg bevacizumab, delivered via intravenous (IV) infusion once every 3 weeks and paclitaxel and carboplatin chemotherapy regimen (paclitaxel 200 mg/m2 and carboplatin at AUC of 6 mg/mL x min) on day 1 of each 3 week cycle for a maximum of 6 cycles.
  Interventions: Biological: Bevacizumab; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Biological: Bevacizumab — 15 mg/kg bevacizumab, delivered via intravenous (IV) infusion once every 3 weeks
  Other Names: Avastin
  Arms: C
Drug: AMG 706 — subjects in Arms A and B will take AMG 706 orally in one of two dosing regimens over each 21-day cycle: •Arm A: 125 mg once daily (QD) •Arm B: 75 mg twice daily every 12 ± approximately 1 hour for 5 days followed by a 2 day treatment free period every 7 days
  Other Names: Motesanib diphosphate
  Arms: A; B
Drug: Paclitaxel — All subjects will receive a paclitaxel chemotherapy regimen (paclitaxel 200 mg/m2) on day 1 of each 3-week cycle for a maximum of 6 cycles.
Drug: Carboplatin — All subjects will receive carboplatin chemotherapy regimen (carboplatin at AUC of 6 mg/mL x min) on day 1 of each 3-week cycle for a maximum of 6 cycles.

SUMMARY:
The purpose of this study is to estimate the difference in objective response rates between each paclitaxel/carboplatin plus AMG 706 arm (Arm A and B) and paclitaxel/carboplatin plus bevacizumab arm (Arm C) in subjects with advanced non-squamous NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18 years or older with histologically or cytologically confirmed advanced non-squamous NSCLC (unresectable stage IIIB with pericardial or pleural effusion or stage IV/recurrent)
* Measureable disease per RECIST criteria modified
* ECOG performance status of 0 or 1
* Ability to take oral medications
* Competent to give written informed consent

Exclusion Criteria:

* Current or prior history of CNS metastases
* Any prior chemotherapy for advanced NSCLC
* History of pulmonary hemorrhage or gross hemoptysis within 6 months prior to randomization
* Prior targeted therapies
* Known history of allergy or hypersensitivity to paclitaxel or carboplatin
* History of arterial or venous thrombosis within 52 weeks prior to randomization
* History of bleeding diathesis or non-pulmonary bleeding within 14 days prior to randomization
* Peripheral neuropathy > grade 1 per CTCAE Version 3.0
* Myocardial infarction, cerebrovascular accident, grade 2 or greater peripheral vascular disease, transient ischemic attack, congestive heart failure, percutaneous transluminal coronary angioplasty/stent, ongoing arrythmias requiring medication or unstable angina within 52 weeks prior to randomization
* Any kind of disorder that compromises the ability of the subject to comply with the study procedures
* Uncontrolled hypertension as defined by resting blood pressure > 150/90 mm Hg. Anti-hypertensive medications are allowed if hypertension is stably controlled at the time of randomization.
* Participation in therapeutic clinical trials or currently receiving other investigational treatment(s) within 30 days prior to randomization
* Pregnant or breast feeding women
* Known to be HIV, hepatitis B surface antigen, or hepatitis C positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2007-01-31 (Actual); Primary Completion 2008-04-23 (Actual); Study Completion 2011-08-03 (Actual)

PRIMARY OUTCOMES:
Objective tumor response rate | Response assessments will be obtained every 6 +/- 1 week until subjects develop disease progression.

SECONDARY OUTCOMES:
Duration of response | Time from first objective tumor response to disease progression or death, if the death was due to disease progression.
Progression free survival | Number of days from randomization tot he date of radiological evidence of disease progression or death.
Overall survival | Time from randomization to death.
Pharmacokinetics of AMG 706 when administered with paclitaxel and carboplatin in Arms A and B | From randomization until disease progression or death.
Safety and tolerability in the 3 arms | From randomization until disease progression or death.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Blumenschein GR Jr, Kabbinavar F, Menon H, Mok TSK, Stephenson J, Beck JT, Lakshmaiah K, Reckamp K, Hei YJ, Kracht K, Sun YN, Sikorski R, Schwartzberg L; Motesanib NSCLC Phase II Study Investigators. A phase II, multicenter, open-label randomized study of motesanib or bevacizumab in combination with paclitaxel and carboplatin for advanced nonsquamous non-small-cell lung cancer. Ann Oncol. 2011 Sep;22(9):2057-2067. doi: 10.1093/annonc/mdq731. Epub 2011 Feb 14. PMID 21321086
- [Background] Claret L, Lu JF, Bruno R, Hsu CP, Hei YJ, Sun YN. Simulations using a drug-disease modeling framework and phase II data predict phase III survival outcome in first-line non-small-cell lung cancer. Clin Pharmacol Ther. 2012 Nov;92(5):631-4. doi: 10.1038/clpt.2012.78. Epub 2012 Aug 22. PMID 22910440
- [Derived] Bass MB, Yao B, Hei YJ, Ye Y, Davis GJ, Davis MT, Kaesdorf BA, Chan SS, Patterson SD. Challenges in developing a validated biomarker for angiogenesis inhibitors: the motesanib experience. PLoS One. 2014 Oct 14;9(10):e108048. doi: 10.1371/journal.pone.0108048. eCollection 2014. PMID 25314641
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com